CLINICAL TRIAL: NCT05663970
Title: Parent-mediated Intervention for Toddlers With Early Social Communication Challenges or Emerging Autism: A Multi-site Randomized Controlled Trial of a Group-based Virtual Program That Empowers Parents as Change Agents
Brief Title: Virtual Group Social ABCs - Multi-site Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: IWK Health Centre (Other); Glenrose Foundation (Other); Dalhousie University (Other); University of Alberta (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Jessica Brian, Clinician Investigator, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0405
Record Dates: First submitted 2022-10-20; First posted 2022-12-23 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder; Social Communication Disorder; Autism or Autistic Traits; Autism Spectrum Disorder With Impaired Functional Language; Autism-Related Speech Delay
MeSH Terms: conditions — Autism Spectrum Disorder; Social Communication Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Group Social ABCs (Experimental): - Participants complete the Group Social ABCs intervention program
  Interventions: Behavioral: VG Social ABCs
- Active Control Condition (No Intervention): * Participants complete the active control condition:
  * 3 bi-weekly (virtual) group-based sessions (i.e., groups of 4-8 parents, over 6 weeks)
  * psychoeducational curriculum not related to social-communication delivered by study personnel not directly involved in the intervention arm
  * Families may access any available services in their communities (i.e., treatment as usual), which are recorded
  * Families will be offered the option to do Group Social ABCs intervention program after completing the Control phase

INTERVENTIONS:
Behavioral: VG Social ABCs — The Social ABCs is an evidence-based caregiver-mediated early intervention. This trial examines the 6-week Virtual Group Social ABCs; an adapted model of the existing evidence-based Social ABCs. The targets are functional directed vocalizations and positive emotion sharing with a caregiver. It is provided to small groups of parents (4-8 per group) who meet virtually for a series of 6 didactic learning sessions led by two trained Coaches, supported by the programs Parent Manual, PowerPoint slides, facilitated discussion, reflection, and idea generation. Each family is assigned a Coach, and one parent per family receives 9 individualized, 1:1 live coaching sessions over a 6-week period via the virtual platform with the goal of learning to implement the Social ABCs strategies with their child. 10-min video recordings of caregiver and child are taken at baseline(time 0), post intervention (time 1),and follow up (time 2) as a measurement of fidelity of implementation and child responsivity.
  Other Names: Social ABCs, Group-based Social ABCs
  Arms: Virtual Group Social ABCs

SUMMARY:
The goal of this randomized control trial is to test the efficacy of the Social ABCs 6 week, group-based model using a virtual delivery platform. The Social ABCs is a caregiver-mediated early intervention program, aiming to increase child skills in directed, intentional vocalizations, and shared smiling with a primary caregiver for toddlers identified as early signs or a confirmed diagnosis of autism spectrum disorder (ASD), or having related social communication challenges. A positive RCT was previously completed using the program's in-person individual, 12-week model, and a pilot study showing preliminary promise of the virtual group-based model has also been published. This adaptation to a virtual, group-based model maintains the core components of the intervention, but allows caregivers to meet and discuss the content as a group from their home environments and complete the program in a shorter timeframe.

The main questions it aims to answer are:

* Is the Social ABCs virtual group-based model an effective early intervention program for toddlers aged 12-42 months with probable or confirmed ASD, or experiencing social communication challenges, when compared to an active control condition?
* Can primary caregivers of these toddlers achieve implementation fidelity in the Social ABCs intervention strategies using the 6-week virtual delivery model? Participants will be randomized into the treatment condition (A) where they will receive the Social ABCs virtual group-based intervention or, into a Control condition (B), where they meet virtually with other caregivers in the control groups over the course of 6 weeks, viewing and discussing 3 didactic presentations around general child development content (not autism- or Social ABCs-specific). Video and questionnaire data will be collected before (Time 0) and after (Time 1) the 6 week period. After an additional 6-8 weeks, the same data will be collected from both groups as a follow-up time point (Time 2).

Researchers will compare the Treatment group and the Control group to measure change in the target behaviours for the child, the caregiver's use of strategies, as well as caregiver stress and self-efficacy, across time-points.

DETAILED DESCRIPTION:
Significant barriers exist to accessing early ASD-specific interventions, including long wait times due to limited system resources (e.g., insufficient funding to meet caseload, lack of sufficient skilled workforce), exacerbated by restrictions to in-person care associated with families' distance from service centres, and now COVID-19 isolation measures.

In response to system pressures and COVID-19 restrictions, the investigators adapted an evidence-based in-person program (the Social ABCs) to increase efficiency and access. Adaptations included (1) abbreviating the duration of the program to 6 (from 12), (2) developing a group-based delivery approach for didactic content, and (3) providing 1:1 coaching over a virtual platform (Zoom for Healthcare). The program builds on an evidence-based in-person model that uses direct in-the-moment coaching to help parents learn skills to support their toddlers' development. The Social ABCs is considered a naturalistic, developmental, behavioural intervention (NDBI), with a focus on child motivation, play-based learning, and shared enjoyment between caregiver and child.

This three-year, multi-site project uses a randomized control trial (RCT) design to evaluate an innovative early intervention program for toddlers with confirmed or suspected autism spectrum disorders (ASD) or related social communication challenges. This study will evaluate whether this innovative virtual group-based approach (VG-Social ABCs) yields child and parent gains compared to an active control condition. The research team will enroll 120 families, recruited from Ontario, Nova Scotia, and Alberta. Toddlers (aged 12 - 42 months), with identified social communication concerns (or a confirmed diagnosis of ASD), and their primary caregiver will be randomized into one of two conditions: (1) VG-Social ABCs or (2) the active control condition. Families randomized into the control condition will have the option to receive the VG-Social ABCs training once their participation in the control phase concludes. Outcome measures include toddler social communication indices and parent implementation fidelity (both derived from video-coding), parent-reported self-efficacy and wellbeing, and child-level social communication outcomes based on parent-report questionnaires.

Analyses will be conducted at the end of the trial. Hypotheses include increased gains (from Time 0 to Time 1) in parent - and child-related variables for families in the Treatment condition, compared to Controls. Investigators also anticipate that child- and parent-related gains will be maintained at Time 2 (i.e., no significant change from Time 1) for the Treatment arm.

The research team developed the virtual model in rapid response to the COVID-19 pandemic, and pilot data shows that this promises to be a powerful way to support families of toddlers with ASD at a developmental stage when they are most amenable to intervention. Beyond COVID-related isolation measures, there continues to be a significant need for increased access to evidence-based early intervention for toddlers with confirmed or probable autism, as many families are currently waiting on years-long waitlists for service. The research team hopes to demonstrate the efficacy of this feasible and resource-efficient intervention to encourage government decision-makers to fund this program for families, leading to increased access to intervention early in life, and improved outcomes for toddlers with ASD and their families. This model will also increase access for families who live in remote and rural regions who often have difficulty accessing important interventions, both within Canada and beyond.

ELIGIBILITY:
Inclusion Criteria:

* ability to comprehend and communicate in English
* access to high-speed internet for virtual participation
* a confirmed diagnosis of ASD made by a qualified professional, or expert clinician impression of red flags for autism spectrum disorder (ASD) or related social communication challenges
* born between 36 and 42 weeks' gestation
* birthweight >2,500g
* no neurological, genetic, or severe sensory or motor conditions
* willing to limit other interventions to 1-hour per week max. if randomized to Treatment Group
* consent to collect video recorded data
* live within the boundaries of clinical supervisors supervision requirements (Ontario, Alberta or Nova Scotia)

Exclusion Criteria:

* failure to meet inclusion criteria

Ages: 12 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Vocal Responsiveness at 6 and 12 Weeks | 12 weeks
  Changes in toddlers' vocal responsiveness to their primary caregivers verbal prompts. Ten minute video recordings coded by blinded research coder in one minute intervals. Data from Baseline (Time 0) compared to data at Week 6 (Time 1) and Week 12 (Time 2).

SECONDARY OUTCOMES:
Change from Baseline Parent Implementation Fidelity at 6 and 12 Weeks | 12 Weeks (Time 0 - Time 1- Time 2)
  Primary caregivers correct use of Social ABCs intervention strategies. Ten minute video recordings coded by blinded research coder in one minute intervals using the 'Social ABCs Parent Fidelity of Implementation Scoring Sheet' (V3, 2021). Successful implementation defined as 75% or higher. Data from Baseline (Time 0) compared to data at Week 6 (Time 1) and Week 12 (Time 2).
Change from Baseline Caregiver Self-Efficacy at 6 and 12 Weeks | 12 Weeks
  Change in caregiver self-reported feelings of empowerment and self-efficacy. Measured using the Parenting Efficacy Measure and the Caregiver Quality of Life Questionnaire, where higher scores indicate higher levels of self-efficacy and feelings of empowerment as a caregiver. Data from Baseline (Time 0) compared to data at Week 6 (Time 1) and Week 12 (Time 2).
Change from Baseline Parent Stress at 6 and 12 Weeks | 12 Weeks
  Change in caregivers self-reported feelings of stress as measured using the Parenting Stress Index, 4th Edition (2012), where higher scores indicate greater stress. Data from Baseline (Time 0) compared to data at Week 6 (Time 1) and Week 12 (Time 2).
Change from Baseline Vocal Initiations at 6 and 12 Weeks | 12 Weeks
  Toddlers' unprompted use of intentional, directed vocalization to primary caregiver. Ten minute video recordings coded by blinded research coder in one minute intervals. Data from Baseline (Time 0) compared to data at Week 6 (Time 1) and Week 12 (Time 2).
Change from Baseline Social Orienting at 6 and 12 Weeks | 12 Weeks
  Toddler socially references primary caregiver unprompted. Ten minute video recordings coded by blinded research coder in one minute intervals. Data from Baseline (Time 0) compared to data at Week 6 (Time 1) and Week 12 (Time 2).
Change in Baseline Words Understood and Used at 6 and 12 Weeks | 12 Weeks
  Change in amount of words understood or used as reported by primary caregiver on the MacArthur-Bates Communicative Development Inventories (CDI), 2nd Edition (2006). Data from Baseline (Time 0) compared to data at Week 6 (Time 1) and Week 12 (Time 2).
Change from Baseline Autism Symptoms at 6 and 12 Weeks | 12 Weeks
  Change in autism or social-communication related skills and challenges as reported by primary caregiver using the PROCESS - Parent Rated Observation of Communication, Emotion, and Social Skills (2006). Data from Baseline (Time 0) compared to data at Week 6 (Time 1) and Week 12 (Time 2).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Brian, PhD, C Psych, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Biggs K, Hind D, Gossage-Worrall R, Sprange K, White D, Wright J, Chatters R, Berry K, Papaioannou D, Bradburn M, Walters SJ, Cooper C. Challenges in the design, planning and implementation of trials evaluating group interventions. Trials. 2020 Jan 29;21(1):116. doi: 10.1186/s13063-019-3807-4. PMID 31996259
- [Background] Brian J, Drmic I, Roncadin C, Dowds E, Shaver C, Smith IM, Zwaigenbaum L, Sacrey LR, Bryson SE. Effectiveness of a parent-mediated intervention for toddlers with autism spectrum disorder: Evidence from a large community implementation. Autism. 2022 Oct;26(7):1882-1897. doi: 10.1177/13623613211068934. Epub 2022 Jan 15. PMID 35037520
- [Background] Brian J, Solish A, Dowds E, Roth I, Bernardi K, Perry K, Daoud S, Jilderda S, MacWilliam S, Smith IM, Zwaigenbaum L, Bryson S. "Going Mobile"-increasing the reach of parent-mediated intervention for toddlers with ASD via group-based and virtual delivery. J Autism Dev Disord. 2022 Dec;52(12):5207-5220. doi: 10.1007/s10803-022-05554-7. Epub 2022 May 24. PMID 35608785
- [Background] Brian JA, Smith IM, Zwaigenbaum L, Bryson SE. Cross-site randomized control trial of the Social ABCs caregiver-mediated intervention for toddlers with autism spectrum disorder. Autism Res. 2017 Oct;10(10):1700-1711. doi: 10.1002/aur.1818. Epub 2017 Jun 2. PMID 28574669
- [Background] Brian JA, Smith IM, Zwaigenbaum L, Roberts W, Bryson SE. The Social ABCs caregiver-mediated intervention for toddlers with autism spectrum disorder: Feasibility, acceptability, and evidence of promise from a multisite study. Autism Res. 2016 Aug;9(8):899-912. doi: 10.1002/aur.1582. Epub 2015 Dec 21. PMID 26688077
- [Background] Penner M, Anagnostou E, Ungar WJ. Practice patterns and determinants of wait time for autism spectrum disorder diagnosis in Canada. Mol Autism. 2018 Mar 6;9:16. doi: 10.1186/s13229-018-0201-0. eCollection 2018. PMID 29541438
- See also: Social ABCs Program Website — https://socialabcs.ca/

DOCUMENTS (1):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT05663970/Prot_000.pdf